CLINICAL TRIAL: NCT07394348
Title: Impact of Biceps Tenotomy Versus Tenodesis on Rehabilitation Outcomes After Rotator Cuff Repair
Brief Title: Impact of Rotator Cuff Repair on Rehabilitation Outcome
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nardin Samuel Nasief, Nardin Samuel Nasief : Principal Investigator, Cairo University
Other Study IDs: Rehab outcomes in Rotator cuff
Record Dates: First submitted 2026-01-26; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Rotator Cuff Repairs
Keywords: Biceps tenotomy; Biceps tenodesis; Rehabilitation outcomes; Hand grip strength

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Biceps tenotomy: Patients will be grouped according to their surgical intervention combined with the rotator cuff repair by orthopaedic surgeon.
  They will be assessed at 3 times interval ( preoperative , within 1 week post operative and after 3 months ).To identify its effect on rehabilitation outcomes in comparison to patients with biceps tenodesis .
  Interventions: Device: Jamar Handheld dynanometer
- Biceps tenodesis: Patients will be grouped according to their surgical intervention combined with the rotator cuff repair by orthopaedic surgeon.
  They will be assessed at 3 times interval ( preoperative , within 1 week post operative and after 3 months ).To identify its effect on rehabilitation outcomes in comparison to patients with biceps tenotomy.
  Interventions: Device: Jamar Handheld dynanometer

INTERVENTIONS:
Device: Jamar Handheld dynanometer — is a precision instrument used to measure isometric grip strength. It is widely recognized in clinical research as the "gold standard" for assessing hand strength and general upper-body physical function due to its high test-retest reliability and inter-instrument validity.

SUMMARY:
This study will investigate the difference between BTT (biceps tenotomy ) versus BTD (biceps tenodesis)in patients undergoing rotator cuff repair on postoperative shoulder pain levels, shoulder function, HGS, forearm supination muscle strength, elbow flexion strength

DETAILED DESCRIPTION:
Rotator cuff tears are common musculoskeletal conditions that are often degenerative and typically affect older adults. They may or may not be symptomatic, and their prevalence increases significantly with age, from approximately 9.7% in individuals under 20 years to 62% in those over 80 years. The rotator cuff plays a critical role in stabilizing the shoulder joint through the concavity-compression mechanism, and its dysfunction can result in shoulder instability, pain, and reduced upper limb strength. Conservative management, including physical therapy, therapeutic modalities, and medications, is considered the first-line approach for treating Rotator cuff tears , while surgical intervention is reserved for cases unresponsive to conservative treatment. Among the commonly performed surgical procedures, biceps tenotomy and biceps tenodesis are often combined with rotator cuff repair to alleviate pain and improve functional outcomes. Hand grip strength is widely recognized as a reliable indicator of overall upper limb function and may be affected by both the pathology and its surgical management. Despite its clinical relevance, limited studies have directly compared the impact of Biceps tenotomy and Biceps tenodesis on Hand grip strength. Furthermore, these surgical techniques may influence other functional outcomes, including elbow flexion strength, forearm supination strength, and pain perception. Therefore, this study seeks to investigate and compare the effects of Biceps tenotomy versus Biceps tenodesis on these parameters in patients undergoing surgical repair for rotator cuff tears.

ELIGIBILITY:
Inclusion Criteria:

The participant's selection will be based on the following criteria:

1. Both genders adults diagnosed with ≥ 1-cm full-thickness tears of rotator cuff.
2. Age ranged from 50 to 70 years .
3. LHB pathology is involved that will receive ARCR combined with biceps tenotomy or tenodesis.
4. Arthroscopically confirmed LHB pathology.
5. Functionality according to their physical level -

Exclusion Criteria:

Participants will be excluded if they have any of the following criteria:

1. Massive irreparable tears.
2. Inflammatory arthritis.
3. Thyroid disease.
4. Glenohumeral osteoarthritis.
5. Severe cervical disorders or paralysis of the axillary nerve.
6. Previous surgery of the affected shoulder.
7. Revision surgeries for a rotator cuff tear.
8. Complete LHBT rupture. -

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 50 all gender patients with rotator cuff tear , they will be selected based on inclusion criteria and allocated based on type of surgery either combined with long head of biceps tenotomy or tenodesis . They will be grouped according to their surgical intervention by orthopaedic surgeon into 2 cohorts .
  25 patients for biceps tenotomy and 25 patients for biceps tenodesis .
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Pain level | 3 time intervals ( pre , within 1 week post , 3 months post )
  Assessed by Visual analog scale : used to assess acute pain particularly effective post-operatively for tracking individual progress .
  The patients mark their current pain level on a 100 mm horizontal line anchored by verbal descriptors .
  Scoring is : 0 for No symptoms , 10 for very severe symptoms
shoulder function | 3 time intervals ( pre , within 1 week post , 3 months post )
  Will be Assessed by Arabic version of American Shoulder and Elbow Suregeons and Constant Score questionnares * American shoulder and Elbow Surgeons used to evaluate shoulder function and pain .
  Patient answer 10 daily activity questions each scored from 0 ( unable) to 3 (normal function ) while the pain assessed by visual analog scale Pain scaore is converted to another 50 point Score total is 100 points ( 50 pain + 50 function ) Higher scores is indication for better shoulder function
  * Constant score used to assess shoulder function recovery . It has 2 sections : 1)subjective : 35 points : patient reports on pain and daily activity ability.
  2)objective : 65 points : clinical measures for range of motion and strength Grading : pain + activities 0_35 points Range of motion +strength 0_65 points Strength is measured as 1 point per pound lifted for 5 sec ..25 points Score total is 100 points .. The higher is better

SECONDARY OUTCOMES:
Hand grip strength | 3 time intervals ( pre , within 1 week post , 3 months post )
  Will be Assessed by jamar handheld dynanometer Three trials of maximum contraction with holding for 3_5 seconds will be conducted .
  The highest value obtained will be used for analysis .
Elbow flexion strength | 3 time intervals ( pre , within 1 week post , 3 months post )
  Will be Assessed by jamar handheld dynanometer Three trials of maximum contraction with holding for 3_5 seconds will be conducted .
  The highest value obtained will be used for analysis .
Forearm supination strength | 3 time intervals ( pre , within 1 week post , 3 months post )
  Will be assessed by jamar handheld dynanometer Three trials of maximum contraction with holding for 3_5 seconds will be conducted .
  The highest value obtained will be used for analysis .

REFERENCES:
- [Background] Liu YC, Huang SW, Adams CR, Lin CY, Chen YP, Kuo YJ, Chuang TY. Preoperative handgrip strength can predict early postoperative shoulder function in patients undergoing arthroscopic rotator cuff repair. J Orthop Surg Res. 2024 Apr 30;19(1):270. doi: 10.1186/s13018-024-04750-8. PMID 38689328
- [Background] Aouad D, El Rassi G. Shoulder Arthroscopic Rotator Cuff Repair With Biceps Tenodesis and Acromioplasty Using a Single Working Portal. Arthrosc Tech. 2021 Mar 22;10(4):e1125-e1129. doi: 10.1016/j.eats.2021.01.005. eCollection 2021 Apr. PMID 33981560